CLINICAL TRIAL: NCT07153666
Title: A Real-world Study on the Influencing Factors of the Efficacy of Ruxolitinib Cream in the Treatment of Vitiligo
Brief Title: A Real-world Study on the Influencing Factors of Efficacy of Ruxolitinib Cream in Vitiligo
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Guo Jin-Zhu, Deputy director of Dermatology Department, Peking University Third Hospital
Other Study IDs: M20250743
Record Dates: First submitted 2025-08-22; First posted 2025-09-04 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Vitiligo
Keywords: vitiligo; JAK; ruxolitinib; treatment; efficacy; influencing factors
MeSH Terms: conditions — Vitiligo | interventions — ruxolitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ruxolitinib: ruxolitinib twice per day
  Interventions: Drug: Ruxolitinib 1.5% Cream BID

INTERVENTIONS:
Drug: Ruxolitinib 1.5% Cream BID — ruxolitinib twice per day

SUMMARY:
Vitiligo is a common chronic autoimmune skin disease that can occur on any part of the body and severely impacts patients' quality of life. Current treatment for vitiligo primarily include topical medications, phototherapy, systemic therapy and surgical interventions, but their efficacy is limited, often failing to achieve ideal therapeutic outcomes, and are associated with a high recurrence rate. This study is an investigator-initiated real-world research on the application of ruxolitinib cream for vitiligo treatment, with the primary objective of exploring the factors influencing the efficacy of ruxolitinib cream in treating vitiligo.

DETAILED DESCRIPTION:
Vitiligo is a common chronic autoimmune skin disease characterized by skin depigmentation, resulting in white patches that can occur on any part of the body and significantly impact patients' quality of life. Currently, treatment options for vitiligo primarily include topical medications, phototherapy, systemic therapy and surgery; however, their efficacy is limited, making it difficult to achieve optimal therapeutic outcomes,with a high recurrence rate. Studies have demonstrated that the JAK-STAT signaling pathway plays a critical role in autoimmune diseases and is involved in the pathogenesis of vitiligo. The JAK inhibitor ruxolitinib cream can improve skin lesions in patients with vitiligo. This study is an investigator-initiated real-world study on the use of ruxolitinib cream for the treatment of vitiligo, with the primary objective of investigating the factors influencing the efficacy of ruxolitinib cream in vitiligo treatment. Primary outcome measure: At Week 24, the clinical characteristic differences between the groups achieving and not achieving T-VASI50 [50% improvement of total vitiligo area scoring index (T-VASI)]. Secondary outcome measures:

(1) At Week 12 and Week 24, the proportion of patients scoring 4(slightly noticeable) or 5(no longer noticeable) on the Vitiligo Noticeability Scale (VNS), as well as the distribution of patients within each category; (2) Change from baseline in vitiligo-specific quality-of-life score (vitiligo-specific quality-of-life, VitiQoL) at Week 12 and Week 24; (3) Proportion achieving T-VASI 50/75/90 at Week 12 and Week 24; (4) Proportion achieving F-VASI 50/75/90[facial vitiligo area scoring index(F-VASI)] at Week 12 and Week24.

ELIGIBILITY:
Inclusion Criteria:

1. Age12 years or older, any gender;
2. Signed"Informed Consent Form";
3. Clinically diagnosed with non-segmental vitiligo;
4. Vitiligo area less than 10% of body surface area;
5. Agreed to discontinue all other vitiligo-related treatments from the screening visit until the final follow-up visit;
6. Female subjects must not plan for pregnancy or oocyte donation from screening until 4 weeks after the last dose and must voluntarily adopt highly effective physical contraception; male subjects must not plan for fertility or sperm donation during the same period and must voluntarily adopt highly effective physical contraception. Methods include:

   * Barrier methods: Condom or barrier cap (diaphragm or cervical cap);
   * Intrauterine device (IUD) or intrauterine system (IUS);
   * Surgical sterilization (bilateral oophorectomy with/without hysterectomy, total hysterectomy, bilateral tubal ligation, or vasectomy) performed ≥6 months prior to the first dose in the subject or their partner;
   * Other investigator-confirmed highly effective physical contraception.

Exclusion Criteria:

1. Allergy to ruxolitinib cream;
2. Pregnant or lactating women;
3. Any condition deemed inappropriate for study participation by the investigator.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: non-segmental vitiligo older than 12 years
Sampling Method: Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
the proportion of achieving T-VASI50 (50% improvement of total vitiligo area scoring index T-VASI) | Week 24
  First, determine the body parts to be evaluated, including the face and neck, palms, upper limbs, trunk, lower limbs and feet, five regions in total. Using the patient's palm as 1% of body surface area to estimate the area of depigmented patches in each body part, measuring the area of depigmented patches within each region. The T-VASI score categorizes the degree of depigmentation into seven levels: 0%, 10%,25%,50%,75%,90%, or 100%. Based on the area of depigmented patches and the degree of depigmentation in each region, the score for each region is calculated according to the T-VASI scoring formula. The specific calculation formula is:T-VASI=∑(number of handprint units occupied by each body part)× the percentage of pigment loss in that region. The score ranges from 0 to 100. The T-VASI50 score represents the proportion of subjects who achieve a≥50% improvement in the Vitiligo Area Scoring Index compared to baseline.

SECONDARY OUTCOMES:
the proportion of patients scoring 4(slightly noticeable) or 5(no longer noticeable) on the Vitiligo Noticeability Scale (VNS) | Week 12 and Week 24
  Vitiligo Noticeability Scale (VNS), a patient-reported outcome measure designed to assess the perceived change in the visibility of facial vitiligo following treatment. Patients are asked to compare the current noticeability of their vitiligo to how it appeared before treatment began. The scale offers five response options, each corresponding to a numerical score:
  More noticeable (score = 1) Equally noticeable (score = 2) Slightly less noticeable (score = 3) Much less noticeable (score = 4) No longer noticeable (score = 5)
Change from baseline in VitiQoL(vitiligo-specific quality-of-life） | Week 12 and Week 24
  Vitiligo-Specific Quality of Life Scale, a comprehensive patient-reported instrument designed to assess the impact of vitiligo on an individual's daily life and well-being over the past month.The scale consists of 16 items. The first 15 items evaluate the frequency and extent of vitiligo's influence across various domains, including emotional state (e.g., feelings of annoyance, embarrassment, depression), social interactions (e.g., worries about others' opinions, difficulty making new friends), daily activities (e.g., clothing choices, grooming, leisure activities), and overall physical health. Patients rate the frequency of each experience on a 7-point Likert scale ranging from 0 ("Not at all") to 6 ("Always"). The final item asks patients to self-assess the overall severity of their skin condition on a similar scale from 0 ("No skin problem") to 6 ("The worst possible case").
Proportion achieving T-VASI 75/90 (75/90% improvement of total vitiligo area scoring index T-VASI) | Week 12 and Week 24
  First, determine the body parts to be evaluated, including the face and neck, palms, upper limbs, trunk, lower limbs and feet, five regions in total. Using the patient's palm as 1% of body surface area to estimate the area of depigmented patches in each body part, measuring the area of depigmented patches within each region. The T-VASI score categorizes the degree of depigmentation into seven levels: 0%, 10%,25%,50%,75%,90%, or 100%. Based on the area of depigmented patches and the degree of depigmentation in each region, the score for each region is calculated according to the T-VASI scoring formula. The specific calculation formula is:T-VASI=∑(number of handprint units occupied by each body part)× the percentage of pigment loss in that region. The score ranges from 0 to 100. The T-VASI 75/90 score represents the proportion of subjects who achieve a≥75/90% improvement in the Vitiligo Area Scoring Index compared to baseline.
Proportion achieving F-VASI 50/75/90(50/75/90% improvement in facial vitiligo area scoring index) | Week 12 and Week24
  The facial Vitiligo Area Scoring Index (F-VASI) range 0 to 3, with higher scores representing a greater area of facial depigmentation across the forehead to original hairline, cheeks to jawline vertically and laterally from corner of mouth to tragus, nose, and eyelids. The F-VASI score categorizes the degree of depigmentation into seven levels: 0%, 10%,25%,50%,75%,90%, or 100%. Based on the area of depigmented patches and the degree of depigmentation in each region, the score for each region is calculated according to the F-VASI scoring formula. The specific calculation formula is: F-VASI=∑(number of handprint units occupied by each body part)× the percentage of pigment loss in that region. The score ranges from 0 to 100. The F-VASI50/75/90 score represents the proportion of subjects who achieve a≥50/75/90% improvement in the Vitiligo Area Scoring Index compared to baseline.

OTHER OUTCOMES:
Safety monitoring-proportion of acne, itching, nasopharyngitis, headache, upper respiratory tract infection, etc. | up to Week 24
  The research doctors inquired about the adverse reactions of the subjects and made records. The subjects reported their own adverse events or reactions.

CONTACTS AND LOCATIONS:
Overall Officials: Jinzhu Guo, MD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No